CLINICAL TRIAL: NCT02086448
Title: Sleep Disordered Breathing, Obesity and Pregnancy Study (SOAP)
Acronym: SOAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francesca Facco, MD (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Francesca Facco, MD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO13080159; R01HL120354 (NIH); K12HD043441 (NIH)
Record Dates: First submitted 2014-02-18; First posted 2014-03-13 (Estimated); Results first posted 2022-03-08 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Obese; Pregnancy; Sleep Disordered Breathing
MeSH Terms: conditions — Obesity; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Obese, SDB negative (No Intervention): No intervention, observational comparison group
- Obese, SDB postive, CPAP (Active Comparator): Therapeutic CPAP
  Interventions: Device: CPAP
- Obese, SDB postive, sham-CPAP (Sham Comparator): Sham (non-therapeutic) CPAP
  Interventions: Device: sham-CPAP
- Obese, SDB postive, sleep hygiene (Other): Sleep hygiene information and local sleep resources
  Interventions: Other: Sleep hygiene

INTERVENTIONS:
Device: CPAP — CPAP is a device that has a mask worn over the nose that is attached to a device that provides positive airway pressure. CPAP is worn while sleeping, it splints open the airway and prevents apneas (cessation of breathing) and hypopneas (reduced airflow while breathing).
  Other Names: Continuous Positive Airway Pressure
  Arms: Obese, SDB postive, CPAP
Device: sham-CPAP
  Arms: Obese, SDB postive, sham-CPAP
Other: Sleep hygiene — Information about sleep apnea and healthy sleep. Information about local sleep resources
  Arms: Obese, SDB postive, sleep hygiene

SUMMARY:
The purpose of this study is to better understand how sleep apnea, a common sleep disorder in which a person has one or more pauses in breathing or shallow breaths while sleeping, may affect pregnancy and to determine the effect of Continuous Positive Airway Pressure (CPAP), a treatment that uses mild air pressure to keep the airways open during sleep, for pregnant women with sleep apnea.

DETAILED DESCRIPTION:
Emerging data support a link between sleep disordered breathing (SDB) and adverse pregnancy outcomes, particularly preeclampsia. Furthermore, SDB, which is characterized by intermittent nocturnal hypoxia-reoxygenation as well as sleep disruption, results in endothelial dysfunction and metabolic dysregulation, the same biological pathways that have been associated with adverse pregnancy outcomes. Obesity is a well-known risk factor for both adverse pregnancy outcomes and SDB, and has been associated with the same aforementioned biological aberrations. Therefore, obesity complicates the definition of a causal relationship between SDB and pregnancy outcomes. While some classic cardiovascular risk factors (prehypertension) are certainly relevant in pregnancy, there are also well-established risk factors that are unique to pregnancy (uterine vascular stiffness, placental angiogenic factors). The interplay between SDB, obesity and these unique cardiovascular risk factors remains undefined, and this proposal aims to address this knowledge gap. Without this data, our ability to understand how we can mitigate these risks through the use of therapeutic interventions for SDB, such as CPAP (continuous positive airway pressure), is compromised. To further address this knowledge gap, we will make use of the placenta's ability to accumulate evidence of damage over time and provide a record of maternal vascular health throughout gestation. Numerous placental lesions deriving from maternal vascular disease have been identified and can be readily detected on placental pathology. These lesions can provide a measure of the severity of hypoxic stress experienced by the fetus during gestation.

The investigators' central hypothesis is that SDB is an effect modifier that increases maternal cardiovascular risk and placental hypoxic injury in obese pregnant women, and that CPAP treatment during pregnancy will result in an improved cardiovascular risk and placental profile. To test this hypothesis the investigaotrs will identify a cohort of obese women both with and without SDB. The investigators will examine SDB's impact on maternal vascular stiffness (uterine artery Doppler), angiogenesis (pregnancy specific angiogenic factors e.g., sFLT-1) and metabolism (insulin resistance) across pregnancy (Aim 1). The investigators will perform a randomized controlled trial of autotitrating- CPAP verses sham-CPAP in pregnancy to examine the impact of CPAP treatment during pregnancy on cardiovascular risk (Aim 2) and will explore the interplay between SDB, CPAP and evidence of maternal vascular disease and chronic fetal hypoxia by evaluating the placental profile of obese women with and without SDB (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* women between 14 0/7 and 20 6/7 weeks gestation at the time of their initial PSG assessment.
* Pregnancy and current BMI >=30
* Self-reported frequent snoring (>=3x/week over past month) or self-reported non-snorer.

Exclusion Criteria:

* diagnosis of pregestational diabetes.
* self-report a history of sleep apena and who are using or were receommended by a physican to use a PAP device already
* twins

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2014-09; Primary Completion 2021-12 (Actual); Study Completion 2022-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Facco, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of the UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Facco FL, Wolsk J, Patel SR, Hubel C, Gallaher M, Cashmere JD, Wisniewski S. A trial of positive airway pressure for the treatment of sleep apnea in pregnancy. Am J Obstet Gynecol MFM. 2023 Mar;5(3):100840. doi: 10.1016/j.ajogmf.2022.100840. Epub 2022 Dec 21. PMID 36563879
- [Derived] Onslow ML, Wolsk J, Wisniewski S, Patel S, Gallaher M, Hubel C, Cashmere DJ, Facco FL. The association between sleep-disordered breathing and maternal endothelial and metabolic markers in pregnancies complicated by obesity. J Clin Sleep Med. 2023 Jan 1;19(1):97-109. doi: 10.5664/jcsm.10254. PMID 36004747

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 452 individuals were screened and 355 participants consented for this study . Prior to or during the inital study visit, 113 individuals withdrew or were withdrawn from the study. 242 participants completed visit 1 (14 0/7-20 6/7 weeks gestation, mean gestational age 18.1 ± 2.0 weeks), of whom 89 (37%) had an AHI between 5 and 50 and therefore were eligible for randomization.
Groups:
- Obese, SDB Postive, CPAP, Phase 1: Therapeutic CPAP
  CPAP: CPAP is a device that has a mask worn over the nose that is attached to a device that provides positive airway pressure. CPAP is worn while sleeping, it splints open the airway and prevents apneas (cessation of breathing) and hypopneas (reduced airflow while breathing).
- Obese, SDB Postive, Sham-CPAP: Sham (non-therapeutic) CPAP
  sham-CPAP
- Obese SDB CPAP Phase 2: Therapeutic CPAP
Period: Overall Study
Arm/Group | Obese, SDB Postive, CPAP, Phase 1 | Obese, SDB Postive, Sham-CPAP | Obese, SDB Postive, Sleep Hygiene | Obese SDB CPAP Phase 2
Started | 25 | 26 | 20 | 18
Completed | 24 | 26 | 20 | 16
Not Completed | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Obese, SDB Positive, CPAP Phase 2: Therapeutic CPAP
- Total: Total of all reporting groups
Arm/Group | Obese, SDB Postive, Sham-CPAP | Obese, SDB Postive, CPAP, Phase 1 | Obese, SDB Postive, Sleep Hygiene | Obese, SDB Positive, CPAP Phase 2 | Total
Number analyzed (Participants) | 26 | 25 | 20 | 18 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (3.9) | 28.4 (6.5) | 32.0 (4.5) | 32.6 (4.5) | 29.6 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 20 | 18 | 89
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 16 | 13 | 9 | 57
  White | 5 | 9 | 6 | 9 | 29
  More than one race | 2 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Uterine Artery Doppler Mean Pulsatility Index -by Ultrasound
Description: The uterine artery was located using color doppler imaging by placing the ultrasound probe in the right or left iliac fossa in the sagittal plane. The uterine artery was then identified where it crosses the external iliac artery. Doppler waveform was obtained using a sampling gate encompassing the width of the main uterine artery at an angle of insonation of <30 degrees if possible. The PI was calculated using the formula: maximum-minimum velocity/mean velocity.
Time Frame: early pregnancy (14-16 weeks gestation)
Measure: Mean (Standard Deviation); unit: Mean PI
Groups:
- Obese, SBD Positive, CPAP, Phase 2: Therapeutic CPAP
Arm/Group | Obese, SDB Postive, Sham-CPAP | Obese, SDB Postive, CPAP, Phase 1 | Obese, SDB Postive, Sleep Hygiene | Obese, SBD Positive, CPAP, Phase 2
Number analyzed (Participants) | 26 | 25 | 20 | 18
Mean PI | 1.0 (0.3) | 1.0 (0.3) | 1.0 (0.3) | 1.0 (0.3)

2. Primary Outcome: Soluble FMS-like Tyrosine Kinase 1 (sFlt-1)/ Placental Growth Factor (PlGF) Ratio-blood Measurement
Description: sFlt-1 is a splice variant of vascular endothelial growth receptor (VEGF) with antiangiogenic properties that is upregulated in preeclampsia. PlGF is an angiogenic cytokine that is highly expressed in the placenta. Low levels have been associated with preeclampsia.
Time Frame: early pregnancy (14-16 weeks gestation)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Obese, SDB Postive, Sham-CPAP | Obese, SDB Postive, CPAP, Phase 1 | Obese, SDB Postive, Sleep Hygiene | Obese, SBD Positive, CPAP, Phase 2
Number analyzed (Participants) | 26 | 25 | 20 | 18
Ratio | 53.8 (29.1) | 65.1 (45.8) | 87.0 (69.1) | 88.3 (45.0)

3. Primary Outcome: Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)-Blood Measurement of Glucose and Insulin
Description: Insulin resistance was calculated using the homeostatic model assessment for insulin resistance (HOMA-IR, fasting insulin (µU/mL) x fasting glucose (mmol/L) /22.5)
Time Frame: early pregnancy (14-16 weeks gestation)
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | Obese, SDB Postive, Sham-CPAP | Obese, SDB Postive, CPAP, Phase 1 | Obese, SDB Postive, Sleep Hygiene | Obese, SBD Positive, CPAP, Phase 2
Number analyzed (Participants) | 26 | 25 | 20 | 18
HOMA-IR score | 4.5 (3.5) | 4.6 (6.4) | 3.9 (2.2) | 4.2 (3.0)

4. Primary Outcome: Uterine Artery Doppler Mean Pulsatility Index -by Ultrasound
Description: as for outcome 1
Time Frame: late pregnancy (28-32 weeks gestation)
Measure: Mean (Standard Deviation); unit: Mean PI
Arm/Group | Obese, SDB Postive, Sham-CPAP | Obese, SDB Postive, CPAP, Phase 1 | Obese, SDB Postive, Sleep Hygiene | Obese, SBD Positive, CPAP, Phase 2
Number analyzed (Participants) | 26 | 24 | 20 | 16
Mean PI | 0.9 (0.2) | 0.8 (0.3) | 0.8 (0.2) | 0.7 (0.1)

5. Primary Outcome: Soluble FMS-like Tyrosine Kinase 1 (sFlt-1)/ Placental Growth Factor (PlGF) Ratio-blood Measurement
Description: as for outcome 2
Time Frame: late pregnancy (28-32 weeks gestation)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Obese, SDB Postive, Sham-CPAP | Obese, SDB Postive, CPAP, Phase 1 | Obese, SDB Postive, Sleep Hygiene | Obese, SBD Positive, CPAP, Phase 2
Number analyzed (Participants) | 26 | 25 | 20 | 18
Ratio | 30.5 (28.9) | 26.0 (18.3) | 38.3 (34.7) | 45.9 (57.3)

6. Primary Outcome: Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)-Blood Measurement of Glucose and Insulin
Description: as for outcome 3
Time Frame: late pregnancy (28-32 weeks gestation)
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | Obese, SDB Postive, Sham-CPAP | Obese, SDB Postive, CPAP, Phase 1 | Obese, SDB Postive, Sleep Hygiene | Obese, SBD Positive, CPAP, Phase 2
Number analyzed (Participants) | 26 | 25 | 20 | 18
HOMA-IR score | 6.3 (10.7) | 3.7 (3.6) | 3.6 (1.8) | 4.6 (6.3)

7. Secondary Outcome: Placental Histology and Immunohistochemistry
Description: placental histology and immunohistochemistry
Time Frame: After delivery (expected 37-40 weeks gestation)
Population: Placental collection and analysis was not performed due to inadequate staffing and personnel issues
Arm/Group | Obese, SDB Postive, Sham-CPAP | Obese, SDB Postive, CPAP, Phase 1 | Obese, SDB Postive, Sleep Hygiene | Obese, SBD Positive, CPAP, Phase 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Other Pre Specified Outcome: Mean Arterial Blood Pressure (mmHg) Angiogenic Domain
Time Frame: early pregnancy (14-16 weeks gestation)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Pregnancy Outcome Data
Description: Preeclampsia, Gestational diabetes, Gestational age at delivery, Indication for delivery, Birthweight, Cord gases
Time Frame: At time of delivery (expected 37-40 weeks gestation)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Mean Arterial Blood Pressure (mmHg) Angiogenic Domain
Time Frame: late pregnancy (28-32 weeks gestation)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Soluble Endoglin (sEng ,pg/mL)-Blood Measurement
Description: Endoglin is a coreceptor for transforming growth factor beta-1 and beta-3 expressed on syncytiotrophoblasts
Time Frame: early pregnancy (14-16 weeks gestation)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Soluble Endoglin (sEng , pg/mL)-Blood Measurement
Description: Endoglin is a coreceptor for transforming growth factor beta-1 and beta-3 expressed on syncytiotrophoblasts
Time Frame: late pregnancy (28-32 weeks gestation)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment to 6 weeks post partum, an average of 1 year
Arm/Group | Obese, SDB Postive, CPAP, Phase 1 | Obese, SDB Postive, Sham-CPAP | Obese, SDB Postive, Sleep Hygiene | Obese, SBD Positive, CPAP, Phase 2
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/26 | 0/20 | 1/18
Other Adverse Events (participants affected / at risk) | 0/25 | 3/26 | 0/20 | 1/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obese, SDB Postive, CPAP, Phase 1 (N=25) | Obese, SDB Postive, Sham-CPAP (N=26) | Obese, SDB Postive, Sleep Hygiene (N=20) | Obese, SBD Positive, CPAP, Phase 2 (N=18)
Maternal ICU admission (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Fetal Demise (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obese, SDB Postive, CPAP, Phase 1 (N=25) | Obese, SDB Postive, Sham-CPAP (N=26) | Obese, SDB Postive, Sleep Hygiene (N=20) | Obese, SBD Positive, CPAP, Phase 2 (N=18)
CPAP complication (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 — When attempting to use the CPAP machine she is waking up in the middle of the night coughing and needing to catch her breath.
EKG abnormality (Cardiac disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT02086448/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT02086448/SAP_001.pdf